CLINICAL TRIAL: NCT03168633
Title: Effects of Reading Information Sent Via Email and Glycemic Control and Compliance to Recommendations Among Patients With Type 2 Diabetes Mellitus -Prospective Research
Brief Title: Lifestyle Advises Sent Via Email in Attempt of Improving A1C in DM2 Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rambam Health Care Campus (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 0456-14-RMB CTIL
Record Dates: First submitted 2017-02-01; First posted 2017-05-30 (Actual); Last update posted 2017-05-30 (Actual); Status verified 2017-05

CONDITIONS: Diabetes Mellitus, Type 2
Keywords: : Type 2 Diabetes Mellitus; Web-based intervention; medication adherence; lifestyle changes
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Medication Adherence

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- patients receiving emails (Experimental): Diagnosed DM2 patients who meet inclusion criteria. the patients will receive emails containing information about DM2 as a method of reminding patients of the importance of adjusting post diagnosis life-style changes.
  web-based DM2 information pages
  Interventions: Behavioral: web-based DM2 information pages

INTERVENTIONS:
Behavioral: web-based DM2 information pages — Each email will include information on one of the following topics:
  1. The importance of physical activity
  2. Correct nutrition
  3. The importance of adhering to medication regimens.
  Emails will be either positive (e.g., the importance of good nutrition, and what constitutes good nutrition) or negative (e.g., the risks of not adhering to medications).
  The information will be provided by different approaches: medical research results, practical tips, patient testimonies.…

SUMMARY:
Diabetic patients need to manage their glucose level, physical activity and food intake to successfully cope with their disease. Previous work has shown that reminders of the disease, be they informational or about ones' condition, can improve management of disease in diabetes.

This trial focuses on delivering these reminders, via email, in attempt to improve the patients glycemic control (measured in Hemoglobin A1C)

DETAILED DESCRIPTION:
The study initially included 50 patients (men and women, over 18 years of age) who were prior diagnosed with DM2 and unbalanced in their glycemic values (HbA1c above 7%). The patient were sent via email , once every other week, a link to web-based pages which provides information on changing DM2 related such as general DM2 information, the importance of keeping a well-balanced diet, benefits of exercising regularly, drug related information and more.

Furthermore, the patients were sent a questionnaire every other week which they were asked to actively reply to.

Each participating patient was monitored for 6 months, during this time he/she was sent 12 web-based information pages.

During the course of the study, information regarding the patients' glycemic control (in the form of HgA1c levels) was collected.

Additional variables (age, sex, BMI, time passed since diagnosed with DM2) were collected and used for statistical comparison.

ELIGIBILITY:
Inclusion Criteria:

1. Previous diabetes specialist follow
2. Age over 18.
3. Diagnosis of diabetes type 2.
4. HbA1c over 7%
5. Self-admitted less than optimal adherence to physical activity, diet or medications or computer-recorded less than 80% adherence to medication purchase.
6. Able to read Hebrew
7. Uses Email account that is actively read at least twice weekly.

Exclusion Criteria:

* Patients who did not the inclusion criteria

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2015-07 (Actual); Primary Completion 2017-01-30 (Actual); Study Completion 2017-01-30 (Actual)

PRIMARY OUTCOMES:
HbA1C values of patients after 6 months | 6 months follow up
  HbA1C values

SECONDARY OUTCOMES:
percentage of messages opened and read | 10-12 messages in 6 months
  reading of each message will be recorded

CONTACTS AND LOCATIONS:
Overall Officials: Irit Hochberg, MD, Principal Investigator — Rambam Hospital

IPD SHARING:
Plan to Share IPD: Undecided